CLINICAL TRIAL: NCT04281329
Title: Contribution of Left Atrial Epicardial Fat Quantification by Computed Tomography and Left Atrial Strain by MRI in Atrial-Fibrilation Ablation: "The CTStrain-AF Study"
Brief Title: Contribution of Computed Tomography and Cardiac-MRI in Atrial Fibrillation Ablation
Acronym: CTStrain-AF
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: University Hospital, Bordeaux (Other); Centre Cardiologique du Nord (Other)
Responsible Party: Sponsor
Other Study IDs: P150925J; N° IDRCB : 2017-A03106-47 (Other: National Agency for the Safety of Medicines)
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Catheter ablation; Magnetic resonance imaging; Computed tomography
MeSH Terms: conditions — Atrial Fibrillation | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Magnetic resonance imaging — Cardiac magnetic resonnance imaging before catheter ablation.

SUMMARY:
Atrial fibrillation ablation (AF) is a standard interventional treatment for patients with symptomatic AF refractory to medical treatment. The known predictive factors for the success of the procedure remain insufficient to predict the probabilities of success and to appropriately select the patients who could benefit the most from this procedure. Left atrium imaging by MRI or CT may be able to identify AF substrate. However data are lacking about the practical impact of these techniques in routine practice to predict AF ablation outcome.

The "CT-AF" study is a prospective, interventional, multicenter cohort study. The main objective of this study is to evaluate the prognostic value of a new automated measurement technique for intra-myocardial atrial fat measurement in cardiac CT and the measurement of global left atrial strain in MRI in patients who are candidates for first AF ablation.

The main outcome will be the relationship between the relative volume of left atrial fat measured with CT and total left atrial strain in MRI and recurrence of AF at 1 year after the ablation procedure (blanking period of 3 months post ablation excluded).

DETAILED DESCRIPTION:
Scientific background :

Atrial fibrillation ablation (AF) is a standard interventional treatment for patients with symptomatic AF refractory to medical treatment. The known predictive factors for the success of the procedure remain insufficient to predict the probabilities of success and to appropriately select the patients who could benefit the most from this invasive procedure. Previous studies have shown that the quantification of atrial fibrosis in magnetic resonance imaging (MRI) may be a good marker of atrial remodeling and would reliably predict the chances of success of the ablation procedure. Nevertheless, the use of this technique is very limited in routine because of the complexity of quantitative analysis and spatial resolution limits. The association of fibrosing processes within epicardial fat has been established. The characterization of epicardial fat in CT could be a relevant substitute for the direct characterization of fibrosis. This examination was essential for the study of atrial anatomy before ablation of AF. In addition to the anatomical evaluation, the study of sub-epicardial fat by cardiac CT could therefore be an interesting approach for evaluating the AF substrate.

Main objective:

To evaluate the prognostic value of a new automated measurement technique for intra-myocardial atrial fat measurement in cardiac CT and the measurement of global left atrial strain in MRI in patients who are candidates for first AF ablation.

Secondary objectives:

* To evaluate the clinical features associated with CT-measured atrial epicardial fat in patients requiring first AF ablation
* To evaluate the clinical features associated with global and regional left atrial strain measured by MRI in patients who are candidates for first AF ablation
* To study global and regional relationships between intramyocardial fat in CT and left atrial strain in MRI
* To evaluate the impact of catheter ablation on the evolution of atrial subepicardial fat measured by CT
* To evaluate the prognostic value of atrial subepicardial fat measured by CT after AF ablation
* To evaluate the relation between subepicardial fat measured by CT and uni-and bipolar voltages mapped in sinus rhythm in patients who are candidates for first AF ablation
* To evaluate the relationship between CT subcuticardic fatness and the distribution of AF-mapped fragmented electrograms in patients who are first-ablated with FA
* To evaluate the relationship between segmental strain measured by MRI and uni and bipolar voltages mapped in sinus rhythm in patients who are candidates for first AF ablation
* To evaluate the relationship between segmental strain measured by MRI and distribution of fragmented electrograms mapped to FA in patients who are candidates for first AF ablation.
* To evaluate the interest of the cartographic fusion function-fat-function-electrophysiology 3D
* To evaluate the relationship between epicardial fat measured by CT and serum biomarkers (adipokines: MMP8 and Activin A, ANF) measured at baseline and at 3 months after ablation
* To evaluate the relationship between segmental strain measured by MRI and serum biomarkers (adipokines: MMP8 and Activin A, ANF) measured at baseline and at 3 months after ablation.

Experimental scheme:

This is a prospective, interventional, multicenter cohort study. Patients with a first radiofrequency or cryotherapy AF ablation are expected to receive a cardiac CT scan (performed for left atrial anatomy study) from which the volume of sub-epicardial fat will be measured. by a new automated measurement technique. The correlation of this measure with the success of ablation (defined as the absence of recurrence of atrial arrhythmia sustained> 30 seconds) will be blinded prospectively to 1 year of follow-up. In addition, the reliability of this measurement will be validated against reference measurements in CT and MRI. The evolution of epicardial fat volume after ablation will be evaluated by a control scan performed as part of the treatment (detection of FA post-ablation pulmonary stenosis). The methods of overall care, imaging examinations and decision criteria at the level of care are common to the 3 investigative centers.

Visits:

V0: selection visit between M-6 and J-1 before ablation (J0)

* Clinical examination, interrogation and antecedents;
* ECG 12D;
* Programming of the preoperative assessment: cardiac scanner after biological assessment with blood ionogram, urea and creatinine and cardiac ultrasound;
* Verification of inclusion and non inclusion criteria;
* Patient information and surrender of consent.

Inclusion visit V1 between the V0 selection visit and the maximum at D-1 before the ablation (J0), after collection of the consent

* Cardiac MRI;
* Biomarker assay and biological collection.
* Recovery of Echocardiography, Standard Biological and Cardiac Scanner data prior to visit V2.

Visit V2: Ablation of FA = J0

* Physical examination ;
* ECG 12D;
* Standard biological assessment;
* Ablation data.

Follow-up visits:

* V3 (M3 +/- 10d): Clinical examination, ECG 12D, holter ECG, cardiac scanner, standard biological assessment, biomarker assay and biological collection.
* V4 (M6 +/- 15d): clinical examination, ECG 12D, holter ECG.
* V5 (M12 +/- 1month) = End of study visit: Clinical examination, ECG 12D, holter ECG.

Number of selected subjects : 130 patients

Number of recruiting centers : 5 centers

ELIGIBILITY:
Inclusion Criteria:

* Patient in whom radiofrequency AF ablation is scheduled within the next 6 months.
* age ≥18 years
* Patient affiliated to a social security scheme
* Patient informed and given written consent for participation in the study.

Exclusion Criteria:

* Refusal to participate in the study
* Patient who has already benefited from an AF ablation procedure
* Patient for whom an AF ablation procedure by cryoablation system is planned
* Scanner or MRI pre-inclusion not exploitable
* Presence of an implantable cardiac prosthesis of pacemaker type or defibrillator
* Claustrophobia
* Iodinated / gadolinium contrast medium allergy
* Chronic renal failure with clearance <30ml / min
* Follow-up visits not possible
* Pregnancy in progress
* Patients unable to sign consent
* Minors and adults protected under legal protection (tutorship or guardianship)
* Period of exclusion from a research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients candidate for a first catheter ablation for atrial fibrillation
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Prognostic value of automated measurement of epicardial fat in CT and and total left atrial strain in MRI | At 1 year
  Relationship between the relative volume of left atrial fat and total left atrial strain in MRI and recurrence of atrial rhythm disturbances (defined as sustained atrial rhythm disturbance> 30 seconds) at 1 year after the ablation procedure (blanking period of 3 months post ablation excluded)

SECONDARY OUTCOMES:
Comparaison of prognostic value of automated measurement of epicardial fat in CT and the references methods | At 1 year
  Comparison of the prognostic value of automated measurement of epicardial fat in CT compared to two reference methods (manual measurement of the reference literature) in all patients .
Comparaison of volume and distribution of left atrial fat and total strail strain with data from electrophysiological mapping | At 1 year
  Global and regional comparison of the relative volume of left atrial fat assessed by CT and left atrial strain assessed by MRI with electroanatomical mapping (voltage and fragmented potential maps) time frame: at one year
Longitudinal study of subepicardial fat volume assessed by CT after ablation | At 1 year
  Comparison of subepicardial left atrial fat volume assessed by CT before and after ablation and prognosis value of the post-ablation subepicardial fat volume on ablation success rate at one year (blanking period of 3 months excluded)
Correlation between the fat volume and the biomarkers. | At 1 year
  The correlation between left atrial fat vollume assessed by CT or left atrial strain assessed by MRI with biomarkers (adipokines: MMP8 and Activin A, ANF) will be studied at baseline and 3 months post ablation. The prognosis value of biomarkers with the ablation success rate at one year (blanking period of 3 months post ablation) will be studied

CONTACTS AND LOCATIONS:
Overall Officials: Alban REDEHEUIL, MD, PhD, Study Director — Centre Hospitalier Universitaire Pitié-Salpêtrière Paris
Locations (1):
- Centre Hospitalier Universitaire Pitie-Salpetriere, Paris, France

REFERENCES:
- [Background] Akoum N, Wilber D, Hindricks G, Jais P, Cates J, Marchlinski F, Kholmovski E, Burgon N, Hu N, Mont L, Deneke T, Duytschaever M, Neumann T, Mansour M, Mahnkopf C, Hutchinson M, Herweg B, Daoud E, Wissner E, Brachmann J, Marrouche NF. MRI Assessment of Ablation-Induced Scarring in Atrial Fibrillation: Analysis from the DECAAF Study. J Cardiovasc Electrophysiol. 2015 May;26(5):473-80. doi: 10.1111/jce.12650. Epub 2015 Apr 23. PMID 25727106
- [Background] Chao TF, Hung CL, Tsao HM, Lin YJ, Yun CH, Lai YH, Chang SL, Lo LW, Hu YF, Tuan TC, Chang HY, Kuo JY, Yeh HI, Wu TJ, Hsieh MH, Yu WC, Chen SA. Epicardial adipose tissue thickness and ablation outcome of atrial fibrillation. PLoS One. 2013 Sep 16;8(9):e74926. doi: 10.1371/journal.pone.0074926. eCollection 2013. PMID 24066158
- [Background] Marrouche NF, Wilber D, Hindricks G, Jais P, Akoum N, Marchlinski F, Kholmovski E, Burgon N, Hu N, Mont L, Deneke T, Duytschaever M, Neumann T, Mansour M, Mahnkopf C, Herweg B, Daoud E, Wissner E, Bansmann P, Brachmann J. Association of atrial tissue fibrosis identified by delayed enhancement MRI and atrial fibrillation catheter ablation: the DECAAF study. JAMA. 2014 Feb 5;311(5):498-506. doi: 10.1001/jama.2014.3. PMID 24496537
- [Background] Samanta R, Pouliopoulos J, Thiagalingam A, Kovoor P. Role of adipose tissue in the pathogenesis of cardiac arrhythmias. Heart Rhythm. 2016 Jan;13(1):311-20. doi: 10.1016/j.hrthm.2015.08.016. Epub 2015 Aug 12. PMID 26277495
- [Background] Venteclef N, Guglielmi V, Balse E, Gaborit B, Cotillard A, Atassi F, Amour J, Leprince P, Dutour A, Clement K, Hatem SN. Human epicardial adipose tissue induces fibrosis of the atrial myocardium through the secretion of adipo-fibrokines. Eur Heart J. 2015 Apr 1;36(13):795-805a. doi: 10.1093/eurheartj/eht099. Epub 2013 Mar 22. PMID 23525094